CLINICAL TRIAL: NCT02226445
Title: Treatment Drop-out and Missed Appointments Among Adults With Attention-Deficit/Hyperactivity Disorder: Associations With Patient- and Disorder-related Factors
Brief Title: Treatment Drop-out and Missed Appointments Among Adults With ADHD
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Sponsor
Other Study IDs: ADHD/DO/MA
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; Drop-out; Non-adherence
Keywords: Adults; Outpatients
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADHD medication and psychosocial counseling
  Interventions: Other: Combined ADHD medication and psychosocial counseling

INTERVENTIONS:
Other: Combined ADHD medication and psychosocial counseling — The patients are offered as well ADHD medication as non-standardized psychosocial treatment, the latter including psychoeducation (i.e. information about ADHD aetiology and symptoms plus management of symptoms) and counselling regarding emotional-, family- and social rehabilitation-related problems.
  ADHD medication:
  First choice of medication is methylphenidate immediate release, initially 5 mg 2-3 times a day increasing with 10-20 mg per week up to stabilization of symptoms.
  When stabilized a shift to extended release methylphenidate. Alternatively dexamphetamine, initially 2.5 mg 2-3 times a day increasing with 5-10 mg per week up to stabilization of symptoms.
  If there is no adequate effect of central stimulants then a shift to atomoxetine, initially 18 mg a day, increasing during a period of 6-10 weeks up to max. 100 mg a day.
  If the patients have a substance use, an anxiety problem or other contraindications then first choice of medication is atomoxetine.

SUMMARY:
The investigators knowledge of factors associated with treatment drop-out and missed appointments among adults with Attention-Deficit/Hyperactivity Disorder (ADHD) within a naturalistic, clinical setting is very limited. Drop-out rates among adult ADHD patients in randomised controlled trials (RCT´s) have been reported to be 26.6% - 50%, and similar rates are reported in two naturalistic studies of medication adherence.

Based on proposed hypotheses that past behaviour patterns are more predictive of current behaviours of treatment drop-out and missed appointments than are sociodemographic and clinical characteristics, the aim of the present study is to examine the associations of 1) sociodemographic variables, 2) clinical variables, 3) risk-taking behaviour 4) educational and occupational instability and 5) behaviours during primary/lower secondary school with treatment drop-out and number of missed appointments.

The target group of the study consists of all patients who initiates assessment at the adult ADHD Clinic at Regional Psychiatric Services West, Herning, Central Denmark Region in the period from September 1, 2010 to September 1, 2011. The patients are referred to this Clinic from general practitioners and specialised psychiatric authorities. The investigators study is designed as an observational, cohort study in which the patients are offered medical and non-manualised psychosocial treatment as it is usually offered in this tertiary ADHD Clinic from which the data are collected.

Data regarding sociodemography, clinical symptoms and impairments, risk-taking behaviour, educational and occupational instability and behaviours during primary/lower secondary school are collected using a semistructured protocol.

In the investigators study the investigators define treatment drop-out as premature termination of ongoing treatment, without any prior clinical or agreed resolution. No standardized definition of treatment drop-out is used through out the literature of adherence to treatment among patients in the psychiatric care system.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the ADHD Clinic and initiating assessment between September 1, 2010 and September 1, 2011

Exclusion Criteria:

* No ADHD diagnosis as assessed by the ADHD Clinic

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients referred to a tertiary ADHD Clinic at Regional Psychiatric Services West, Central Denmark Region
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Treatment drop-out | Patients will be followed for the duration of outpatient treatment at the ADHD Clinic, an expected average of 1 year
  The outcome measure "treatment drop-out" is a binary outcome where participants at discharge are characterized as "drop-outs" or "non drop-outs".
  "Drop-outs" are defined as those participants, who terminate treatment without any prior clinical or agreed resolution.
  Logistic regression analyses is applied to calculate outcome odds ratios.
Missed appointments | Patients will be followed for the duration of outpatient treatment at the ADHD Clinic, an expected average of 1 year
  The outcome measure "missed appointments" is a binary outcome, dichomized into <3 missed appointments during treatment and ≥3 missed appointments during treatment.
  Logistic regression analyses is applied to calculate outcome odds ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Jørgen Søgaard, MD, Ph.d., Study Chair — Psychiatric Research Unit West, Regional Psychiatric Services West, Central Denmark Region; Helle Møller Søndergaard, MSc, Principal Investigator — Psychiatric Research Unit West, Regional Psychiatric Services West, Central Denmark Region; Per Hove Thomsen, Professor, Study Chair — Center for Child and Adolescent Psychiatry, Aarhus University Hospital, Central Denmark Region; Erik Pedersen, MD, Study Chair — Regional Psychiatric Services West, Central Denmark Region
Locations (1):
- Psychiatric Research Unit West, Regional Psychiatric Services West, Herning, Denmark

REFERENCES:
- [Derived] Soendergaard HM, Thomsen PH, Pedersen P, Pedersen E, Poulsen AE, Nielsen JM, Winther L, Henriksen A, Rungoe B, Soegaard HJ. Treatment dropout and missed appointments among adults with attention-deficit/hyperactivity disorder: associations with patient- and disorder-related factors. J Clin Psychiatry. 2016 Feb;77(2):232-9. doi: 10.4088/JCP.14m09270. PMID 26761266